CLINICAL TRIAL: NCT03144583
Title: Pilot Study on the Infusion of Differentiated Autologous T-cells From Peripheral Blood, Expanded and Transduced With a Lentivirus to Express a Chimeric Antigen Receptor With Anti-CD19 Specificity Conjugated With the Co-stimulatory Regions 4-1BB and CD3z in Patients With CD19+ Leukemia or Lymphoma Refractory to Therapy
Brief Title: Pilot Study on the Infusion of ARI-0001 Cells in Patients With CD19+ Leukemia or Lymphoma Refractory to Therapy
Acronym: CART19-BE-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sara V. Latorre (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Sara V. Latorre, Clinical Research Manager, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Organization: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CART19-BE-01
Record Dates: First submitted 2017-04-26; First posted 2017-05-09 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Leukemia; Lymphoma
Keywords: CART19
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult differentiated autologous T-cells (Experimental): Adult differentiated autologous T-cells from peripheral blood, expanded and transduced with a lentivirus to express a chimeric antigen receptor with anti-CD19 specificity (A3B1) conjugated with the co-stimulatory regions 4-1BB and CD3z. Such cells will be administered in a single infusion intravenously at a total ARI-0001 cell dose of 0.5-10 x 106 / kg body weight.
  Interventions: Biological: Adult differentiated autologous T-cells

INTERVENTIONS:
Biological: Adult differentiated autologous T-cells — After pretreatment, adult differentiated autologous T-cells with a chimeric antigen receptor with anti-CD19 specificity will be transfused.

SUMMARY:
To assess the infusion of ARI-0001 cells (Adult differentiated autologous T-cells from peripheral blood, expanded and transduced with a lentivirus to express a chimeric antigen receptor with anti-CD19 specificity [A3B1] conjugated with the co-stimulatory regions 4-1BB and CD3z ) safety on patients with leukemia or lymphoma CD19+ resistant or refractory to treatment and with a prognosis of less than 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of leukemia or CD19 + lymphoma, with a life expectancy less than 2 years that meet the following conditions:- Adult acute lymphoid leukemia in second or third response, not candidate for transplantation due to age, associated diseases or lack of donor, or in relapse post allogeneic transplant.- Pediatric acute lymphoid leukemia in second or third response, refractory or non-transplant candidate due to donor absence, or in relapse post allogeneic transplant, or with minimal residual residual disease (0.1% or greater) after two or more lines of treatment. - Symptomatic follicular lymphoma, which has received at least 2 treatment regimens (one of them including rituximab) and a progression-free interval of less than 2 years. Patients not candidates for transplantation or post-transplant relapse may be included.- Symptomatic chronic lymphocytic leukemia, which has received at least 2 treatment regimens (one of them including rituximab) and a progression-free survival of less than 2 years. Patients with a 17p deletion or TP53 mutation may be included after the first line of treatment. - Mantle cell lymphoma in the first relapse (or higher) when it is not a candidate for transplantation, or second post-transplant relapse (or higher). - Diffuse large cell lymphoma in first relapse (or higher) when it is not a candidate for transplantation, or second post-transplant relapse (or higher).
* Age greater than 2 years and less than 80.
* ECOG functional status from 0 to 2
* Life expectancy of at least 3 months.
* Appropriate venous access to perform an apheresis procedure. Absence of contraindications for it.
* Signature of informed consent (patient or legal guardian).

Exclusion Criteria:

* Treatment with any experimental or non-marketed substance within four weeks prior to recruitment, or actively participating in another therapeutic clinical trial.
* Diagnosis of another past or present neoplasm. Patients may be included in complete remission for more than 3 years, or with a history of non-melanoma skin cancer or completely resected in-situ carcinoma.
* Central nervous system involvement (CNS-3) at inclusion. Inclusion will be permitted with patients with a lower grade (CNS-2) or with CNS-3 who have responded to intrathecal chemotherapy.
* Early relapse after allogeneic transplantation (less than 3 months for apheresis of mononuclear cells, less than 6 months for infusion of ARI-0001) or patients on active immunosuppressive therapy for graft-versus-host disease (corticosteroids or other systemic immunosuppressants ).
* Active infection requiring systemic medical treatment such as chronic kidney infection, chronic lung infection or tuberculosis.
* HIV infection.
* Concurrent and uncontrolled medical illnesses including cardiac, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological or psychiatric diseases which in the opinion of the researcher represent a risk to the patient.
* Positive serology for hepatitis B, defined as a positive test for HBsAg. In addition, if the patient is HBsAg negative but has anti-HBc antibodies it will be necessary to perform a DNA test of the hepatitis B virus, and if the result is positive the patient will be excluded.
* Positive serology for hepatitis C, defined as a positive test for anti-HCV antibodies confirmed by RIBA.
* Severe organ failure, defined as a cardiac ejection fraction <40%; DLCO <40%; calculated glomerular filtrate rate <30 ml / min; Or bilirubin> 3 times the upper limit of normal (unless it is due to CLL or Gilbert syndrome).
* Pregnant or lactating women. Women of childbearing potential should have a negative pregnancy test in the screening phase.
* Women of childbearing age, including those whose last menstrual cycle was in the year prior to screening, who are unable or unwilling to use highly effective contraceptive methods from the start of the study to the end of the study.
* Men who are unable or unwilling to use highly effective contraceptive methods from the start of the study to the completion of the study.
* The need to take glucocorticoids in a chronic manner at doses higher than 10 mg / day of prednisone (or equivalent) or other chronic immunosuppressants. Hormonal contraceptives, intrauterine device, intrauterine systems of hormonal release, sexual abstinence, vasectomy of the couple or bilateral tubal occlusion.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Procedure-related mortality (PRM) | Year 1
  Any death not caused directly by leukemia / lymphoma. For the estimation of PRM, relapse or progression of the disease will be considered as a competitive event.
Procedure-related mortality (PRM) | Year 3
  Any death not caused directly by leukemia / lymphoma. For the estimation of PRM, relapse or progression of the disease will be considered as a competitive event.
Assessment of toxicity | Month 3
  number of adverse events grade III-IV using CTC (common toxicity criteria)
Assessment of toxicity | Year 1
  number of adverse events grade III-IV using CTC (common toxicity criteria)

SECONDARY OUTCOMES:
Response rate (overall and complete) | Month 3 and Year 1
  Defined differently for each disease:
  * On chronic lymphoid and acute lymphocytic leukemia, the usual criteria NCCN and IWCLL will be used.
  * On non-Hodgkin's lymphoma, the Lugano criteria will be used-
  * On patients with leukemia will be quantified the persistence of minimal residual disease, in bone marrow and peripheral blood, using multiparametric cytometry and new generation sequencing techniques.
Progression-free survival | Year 2 after procedure
  Time lag between infusion of ARI-0001 and the progression of disease or death. Patients alive and in complete remission will be censored at the last follow-up
Overall survival (OS) at 2 years | 3 years
  Time lag between the infusion of ARI-0001 and the death of the patient from any cause. Living patients will be censored at the the last follow-up.
In vivo survival of ARI-0001 cells in peripheral blood, bone marrow and cerebrospinal fluid | months 1,2,3,4,5,6
  Determined monthly during the first 6 months by flow cytometry and quantitative transgene PCR.
In vivo survival of ARI-0001 cells in peripheral blood, bone marrow and cerebrospinal fluid | months 9,12,15,18,21,24
  Determined quarterly from month 6 until the 2 years after infusion, by flow cytometry and quantitative transgene PCR.
Quality of life of included patients | Month 3, 6, 12
  Evaluated by a questionnaire completed by patients or their legal guardians
Toxicity assessment | Month 3 and year 1
  defined as number of adverse events of any type occurring throughout the study using the common toxicity criteria

CONTACTS AND LOCATIONS:
Overall Officials: Julio Delgado González, PhD MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (2):
- Spain (2):
  - Hospital Clínic of Barcelona, Barcelona
  - Hospital Sant Joan de Deu, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bartolo-Ibars A, Aran A, Johansson AM, Ortiz-Maldonado V, Klein-Gonzalez N, Alonso-Saladrigues A, James E, Urbano-Ispizua A, Rives S, Delgado J, Gonzalez-Navarro EA, Kwok WW, Juan M. T-cell responses against CD19-targeted CAR T cells varnimcabtagene autoleucel (ARI-0001): implications for immune response and therapy outcomes. J Immunother Cancer. 2025 Sep 22;13(9):e010792. doi: 10.1136/jitc-2024-010792. PMID 40987492
- [Derived] Martinez-Cibrian N, Ortiz-Maldonado V, Espanol-Rego M, Alserawan L, Navarro S, Albiol N, Lozano M, Charry P, Magnano L, Rivero A, Correa JG, Mozas P, Cortes-Bullich A, Jimenez-Vicente C, Gine E, Montoro-Lorite M, Ramos C, Ayora P, Calderon H, Sanchez-Castanon M, Benitez-Ribas D, Mata-Molanes JJ, Rojas K, Setoain X, Rodriguez S, Murias A, Alcubilla P, Varea S, Olesti E, Bachiller M, Calvo-Orteu M, Sans-Pola C, Saez-Penataro J, de Larrea CF, Lopez-Guillermo A, Gonzalez-Navarro EA, Juan M, Delgado J. Efficacy and safety of the academic anti-CD19 chimeric antigen receptor T-cell product varnimcabtagene autoleucel for the treatment of relapsed/refractory follicular lymphoma. Hemasphere. 2025 Sep 11;9(9):e70166. doi: 10.1002/hem3.70166. eCollection 2025 Sep. PMID 40951523
- [Derived] Martinez-Cibrian N, Ortiz-Maldonado V, Espanol-Rego M, Blazquez A, Cid J, Lozano M, Magnano L, Gine E, Correa JG, Mozas P, Rodriguez-Lobato LG, Rivero A, Montoro-Lorite M, Ayora P, Navarro S, Alserawan L, Gonzalez-Navarro EA, Castella M, Sanchez-Castanon M, Cabezon R, Benitez-Ribas D, Setoain X, Rodriguez S, Brillembourg H, Varea S, Olesti E, Guillen E, Saez-Penataro J, de Larrea CF, Lopez-Guillermo A, Pascal M, Urbano-Ispizua A, Juan M, Delgado J. The academic point-of-care anti-CD19 chimeric antigen receptor T-cell product varnimcabtagene autoleucel (ARI-0001 cells) shows efficacy and safety in the treatment of relapsed/refractory B-cell non-Hodgkin lymphoma. Br J Haematol. 2024 Feb;204(2):525-533. doi: 10.1111/bjh.19170. Epub 2023 Oct 31. PMID 37905734
- [Derived] Ortiz-Maldonado V, Rives S, Castella M, Alonso-Saladrigues A, Benitez-Ribas D, Caballero-Banos M, Baumann T, Cid J, Garcia-Rey E, Llanos C, Torrebadell M, Villamor N, Gine E, Diaz-Beya M, Guardia L, Montoro M, Catala A, Faura A, Gonzalez EA, Espanol-Rego M, Klein-Gonzalez N, Alsina L, Castro P, Jordan I, Fernandez S, Ramos F, Sune G, Perpina U, Canals JM, Lozano M, Trias E, Scalise A, Varea S, Saez-Penataro J, Torres F, Calvo G, Esteve J, Urbano-Ispizua A, Juan M, Delgado J. CART19-BE-01: A Multicenter Trial of ARI-0001 Cell Therapy in Patients with CD19+ Relapsed/Refractory Malignancies. Mol Ther. 2021 Feb 3;29(2):636-644. doi: 10.1016/j.ymthe.2020.09.027. Epub 2020 Sep 20. PMID 33010231
- [Derived] Castella M, Caballero-Banos M, Ortiz-Maldonado V, Gonzalez-Navarro EA, Sune G, Antonana-Vidosola A, Boronat A, Marzal B, Millan L, Martin-Antonio B, Cid J, Lozano M, Garcia E, Tabera J, Trias E, Perpina U, Canals JM, Baumann T, Benitez-Ribas D, Campo E, Yague J, Urbano-Ispizua A, Rives S, Delgado J, Juan M. Point-Of-Care CAR T-Cell Production (ARI-0001) Using a Closed Semi-automatic Bioreactor: Experience From an Academic Phase I Clinical Trial. Front Immunol. 2020 Mar 20;11:482. doi: 10.3389/fimmu.2020.00482. eCollection 2020. PMID 32528460